CLINICAL TRIAL: NCT01116648
Title: Phase I/II Study of Cediranib and Olaparib in Combination for Treatment of Recurrent Papillary-Serous Ovarian, Fallopian Tube, or Peritoneal Cancer or for Treatment of Recurrent Triple-Negative Breast Cancer
Brief Title: Cediranib Maleate and Olaparib in Treating Patients With Recurrent Ovarian, Fallopian Tube, or Peritoneal Cancer or Recurrent Triple-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02938; NCI-2012-02938 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2010-01329; DFCI IRB 09-293; NCI-2013-00578; 8348 (Other: Dana-Farber Cancer Institute); 8348 (Other: CTEP); N01CM00071 (NIH); P30CA006516 (NIH); U01CA062490 (NIH); UM1CA186709 (NIH); NCT01115829 (obsolete NCT alias)
Record Dates: First submitted 2010-04-29; First posted 2010-05-05 (Estimated); Results first posted 2020-07-22 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Fallopian Tube Carcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian High Grade Serous Adenocarcinoma; Ovarian Serous Adenocarcinoma; Ovarian Serous Surface Papillary Adenocarcinoma; Primary Peritoneal Serous Adenocarcinoma; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Triple Negative Breast Neoplasms | interventions — Biopsy; Specimen Handling; cediranib; Magnetic Resonance Spectroscopy; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (cediranib maleate and olaparib) (Experimental): Patients receive cediranib maleate PO QD and olaparib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo CT or MRI as well as blood sample collection on the trial. Patients may also optionally undergo a tissue biopsy on the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Olaparib
- Arm II (olaparib) (Active Comparator): Patients receive olaparib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo CT or MRI as well as blood sample collection on the trial. Patients may also optionally undergo a tissue biopsy on the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Olaparib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo optional tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
  Arms: Arm I (cediranib maleate and olaparib)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281

SUMMARY:
This partially randomized phase I/II trial studies the side effects and the best dose of cediranib maleate and olaparib and to see how well they work compared to olaparib alone in treating patients with ovarian, fallopian tube, peritoneal, or triple-negative breast cancer that has returned after a period of improvement (recurrent). Cediranib maleate may help keep cancer cells from growing by affecting their blood supply. Olaparib may stop cancer cells from growing abnormally. The combination of cediranib maleate and olaparib may be safe, tolerable and/or effective in treating patients with recurrent ovarian, fallopian tube, or peritoneal cancer or recurrent triple-negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the maximum tolerated dose (MTD) of cediranib maleate (cediranib) in combination with olaparib in the treatment of recurrent ovarian, fallopian tube, or peritoneal cancer or metastatic triple-negative breast cancer. (Phase I) II. Assess the efficacy (as measured by progression-free survival [PFS]) of the combination of cediranib and olaparib compared to olaparib alone in recurrent grade 2 or 3 platinum-sensitive papillary-serous or endometrioid ovarian, fallopian tube, or peritoneal cancer. (Phase II) III. Assess the MTD of cediranib in combination with olaparib tablet formulation in the treatment of recurrent ovarian, fallopian tube, or peritoneal cancer. (Phase I-T) IV. Assess the toxicities of the combination of cediranib and olaparib (tablet formulation) in the treatment of recurrent ovarian, fallopian tube, or peritoneal cancer. (Phase I-T) V. Assess clinical benefit, progression-free survival, and overall survival for patients treated with cediranib and olaparib (tablet formulation). (Phase I-T) VI. Assess the pharmacokinetic profile of cediranib and olaparib (tablet formulation) when administered in combination. (Phase I-T)

SECONDARY OBJECTIVES:

I. Assess the toxicities of the combination of cediranib and olaparib in the treatment of recurrent ovarian, fallopian tube, or peritoneal cancer or metastatic triple-negative breast cancer. (Phase I) II. Assess clinical benefit, progression-free survival, and overall survival for patients treated with cediranib and olaparib. (Phase I) III. Assess tumor response, clinical response benefit (response or stable disease as defined by Response Evaluation Criteria in Solid Tumors [RECIST] response criteria x 16 weeks), and overall survival (OS) for patients treated with cediranib and olaparib at the recommended phase II dose (RP2D) as compared with patients receiving olaparib alone. (Phase II)

TRANSLATIONAL OBJECTIVES:

I. To evaluate the prognostic and predictive role of measured changes in functional vascular imaging using dynamic contrast-enhanced (DCE)-magnetic resonance imaging (MRI) between pre-study and day 3. (Phase II) II. To evaluate in an exploratory fashion the predictive or prognostic value of single nucleotide polymorphisms (SNPs) in key genes involved in angiogenesis and deoxyribonucleic acid (DNA) repair. (Phase II) III. To evaluate the predictive value of baseline peripheral blood mononuclear cells (PBMC) poly adenosine diphosphate (ADP) ribose (PAR) incorporation on response to therapy. (Phase II) IV. To measure early changes in vascular cytokine production and evaluate in an exploratory fashion that these changes may be predictive or prognostic, or differentially affected by the combination of agents. (Phase II) V. To evaluate early changes to circulating endothelial cells and if these changes are predictive or prognostic. (Phase II) VI. To assess changes in measures of DNA damage and repair and angiogenesis in tumor cells (tissue and/or malignant effusions) and correlate to drug/drug/combination. (Phase II)

OUTLINE: This is a phase I, dose-escalation study followed by a randomized phase II study.

PHASE I: Patients receive cediranib maleate orally (PO) once daily (QD) and olaparib PO twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening and as clinically indicated on study. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) as well as blood sample collection on the trial. Patients may also optionally undergo a tissue biopsy on the trial.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cediranib maleate PO QD and olaparib PO BID on days 1-28.

ARM II: Patients receive olaparib PO BID on days 1-28.

In both arms, cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening and as clinically indicated on study. Patients also undergo CT or MRI as well as blood sample collection on the trial. Patients may also optionally undergo a tissue biopsy on the trial.

After completion of study treatment, patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I: Participants must have histologically or cytologically confirmed epithelial ovarian cancer, primary peritoneal serous cancer, fallopian tube cancer, or triple-negative breast cancer
* PHASE II: Participants must have histologically or cytologically grade 2 or 3 (high-grade) papillary-serous or endometrioid epithelial ovarian cancer, primary peritoneal serous cancer, or fallopian tube cancer; participants with epithelial ovarian, primary peritoneal, or fallopian tube cancers of other high-grade histologies who carry a known deleterious breast cancer gene (BRCA) germline mutation by standard clinical testing (Myriad BRAC Analysis) will also be considered eligible
* PHASE I-T: Participants must have histologically or cytologically confirmed epithelial ovarian cancer, primary peritoneal serous cancer, or fallopian tube cancer
* Ovarian cancer, primary peritoneal, and fallopian tube participants in the Phase 1 and Phase 1-T portions of this trial must have either measurable cancer by RECIST 1.1 criteria or an elevated cancer antigen (CA)125 level at least twice the upper limit of normal on two separate occasions at least 1 day but not more than 3 months apart; at least one of the samples should be within 1 week of starting treatment; patients with both an elevated CA125 and measurable cancer will be followed by RECIST 1.1 criteria; patients with only an elevated CA125 level will be followed by modified Gynecologic Cancer Intergroup (GCIG) criteria
* Participants in the Phase II portion of the trial must have measurable disease by RECIST 1.1 criteria
* Breast cancer participants must have measurable disease by RECIST criteria
* PRIOR THERAPY PHASE I and PHASE I-T:

  * Prior chemotherapy for ovarian cancer patients must have included a first-line platinum-based regimen with or without intravenous consolidation chemotherapy
  * Breast cancer patients must have recurred post both an Adriamycin- and taxane-containing regimen
  * Prior hormonal-based therapy for ovarian, primary peritoneal serous, fallopian tube cancer, or breast cancer is acceptable
  * Patients may not have had a prior PAR polymerase (PARP)-inhibitor in the recurrent or metastatic setting; prior treatment with BSI-201 (iniparib) is allowed
  * Patients may not have had a prior anti-angiogenic agent in the recurrent or metastatic setting
* PRIOR THERAPY PHASE II:

  * Prior chemotherapy must have included a first-line platinum-based regimen with or without intravenous consolidation chemotherapy
  * Prior hormonal-based therapy for ovarian, primary peritoneal serous, or fallopian tube cancer is acceptable
  * Patients may not have previously received a PARP-inhibitor; prior treatment with BSI-201 is allowed
  * Patients may not have had a prior anti-angiogenic agent in the recurrent setting
  * Patients may have received up to 1 non-platinum-based line of therapy in the recurrent setting
  * Patients may have received an unlimited number of platinum-based therapies in the recurrent setting
  * Patients should have platinum-sensitive disease, where platinum-sensitive disease is defined as having had a > 6 month interval since last receiving platinum therapy prior to disease recurrence; patients must have had a prior response while on the platinum-containing regimen and cannot have experienced disease progression while receiving platinum
* Subjects may begin cediranib and olaparib at least 3 weeks after their last dose of chemotherapy or hormonal therapy, assuming they are otherwise eligible
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of cediranib or olaparib in participants < 18 years of age, children are excluded from this study but will be eligible for future pediatric trials
* Estimated life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky > 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin > 9 g/dL

  * For patients enrolled to the Phase 1-T portion of the protocol, the hemoglobin should be >= 10 g/dL
* Total bilirubin within 1.5 times the upper limit of normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine =< the institutional upper limit of normal or creatinine clearance >= 60 mL/min/1.73 m^2 for subjects with creatinine levels above institutional normal
* Less than or equal to 1+ proteinuria on two consecutive dipsticks taken no less than 1 week apart, or < 1 gm protein on 24-hour urine collection or a urine protein: creatinine ratio of < 1
* Troponin T or I within normal institutional limits
* Coagulation parameters (international normalized ratio [INR], activated partial thromboplastin time [aPTT]) within 1.25 x upper limit of normal institutional limits, except where a Lupus anti-coagulant has been confirmed
* Toxicities of prior therapy (except alopecia) should be resolved to less than or equal to grade 1 as per National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (NCI-CTCAE v4.0); patients with long-standing stable grade 2 neuropathy may be considered after discussion with the overall principal investigator (PI)
* Subjects with treated limited stage basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the breast or cervix are eligible; subjects with prior cancer treated with a curative intent with no evidence of recurrent disease 5 years following diagnosis and judged by the investigator to be at low risk of recurrence are eligible; subjects with any other concomitant or prior invasive malignancies are ineligible
* Patients who have the following risk factors are considered to be at increased risk for cardiac toxicities; these patients should have increased monitoring:

  * Prior treatment with anthracyclines
  * Prior treatment with trastuzumab
  * A New York Heart Association classification of II controlled with treatment
  * Prior central thoracic radiation therapy (RT), including RT to the heart
  * History of myocardial infarction within 12 months (patients with history of myocardial infarction within 6 months are excluded from the study)
* The effects of cediranib and olaparib on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 3 months following treatment discontinuation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent
* Patients must be able to tolerate oral medications and not have gastrointestinal illnesses that would preclude absorption of cediranib or olaparib
* Patients must be willing and able to check and record daily blood pressure readings

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier
* Participants may not be receiving any other investigational agents nor have participated in an investigational trial within the past 4 weeks; subjects may not have received prior treatment affecting the vascular endothelial growth factor (VEGF) pathway in the recurrent setting, including thalidomide, bevacizumab, sunitinib, or sorafenib; in the Phase I portion of the trial, subjects may not have received prior treatment with oregovomab (OvaRex) or any other antibodies that may interfere with CA-125 measurements
* Patients with untreated brain metastases, spinal cord compression, or evidence of symptomatic brain metastases or leptomeningeal disease as noted on computed tomography (CT) or MRI scans should not be included on this study, since neurologic dysfunction may confound the evaluation of neurologic and other adverse events; screening imaging to rule out brain metastases is not required for screening, but should be performed prior to study enrollment if clinically indicated; patients with treated brain metastases and resolution of any associated symptoms must demonstrate stable post-therapeutic imaging for at least 6 months following therapy prior to starting study drug
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cediranib maleate or olaparib
* Participants receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) are ineligible; dihydropyridine calcium-channel blockers are permitted for management of hypertension
* Patients with any of the following:

  * History of myocardial infarction within six months
  * Patients with corrected QT (QTc) prolongation > 500 msec or other significant electrocardiogram (ECG) abnormality noted within 14 days of treatment

    * For patients enrolled in the Phase 1-T portion of the protocol, the QTc should not exceed 470 msec
  * New York Heart Association (NYHA) classification of III or IV
  * If cardiac function assessment is clinically indicated or performed: left ventricular ejection fraction (LVEF) less than normal per institutional guidelines, or < 55%, if threshold for normal not otherwise specified by institutional guidelines
  * Condition requiring concurrent use of drugs or biologics with pro-arrhythmic potential
* History of stroke or transient ischemic attack within six months
* Patients may not have any evidence of pre-existing inadequately controlled hypertension (defined as a systolic blood pressure [BP] of > 140 mmHg or a diastolic BP of > 90 mmHg), and must have a normal blood pressure (=< 140/90 mmHg) taken in the clinic setting by a medical professional within 2 weeks prior to starting study; patients with hypertension may be managed with up to a maximum of three antihypertensive medications; patients who are on three antihypertensive medications must be actively followed by a cardiologist or blood pressure specialist for management of blood pressure while on protocol
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Clinical significant peripheral vascular disease or vascular disease (aortic aneurysm or aortic dissection)
* Unstable angina
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting cediranib
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess
* Current signs and/or symptoms of bowel obstruction or signs and/or symptoms of bowel obstruction within 3 months prior to starting study drugs
* Current dependency on intravenous (IV) hydration or total parenteral nutrition (TPN)
* Evidence of coagulopathy or bleeding diathesis; therapeutic anticoagulation for prior thromboembolic events is permitted
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because cediranib and olaparib are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with cediranib and olaparib, breastfeeding should be discontinued if the mother is treated with cediranib or olaparib; these potential risks may also apply to other agents used in this study
* Known human immunodeficiency virus (HIV)-positive individuals are ineligible because of the potential for pharmacokinetic interactions with cediranib or olaparib; in addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Patients may not use natural herbal products or other "folk remedies" while participating in this study
* No features suggestive of myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML) on peripheral blood smear or bone marrow biopsy, if clinically indicated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2010-04-14 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2026-02-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce F Liu, Principal Investigator — Dana-Farber Cancer Institute
Locations (14):
- United States (14):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc - Jefferson Boulevard, Fort Wayne, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - National Cancer Institute, Rockville, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Liu JF, Barry WT, Birrer M, Lee JM, Buckanovich RJ, Fleming GF, Rimel B, Buss MK, Nattam S, Hurteau J, Luo W, Quy P, Whalen C, Obermayer L, Lee H, Winer EP, Kohn EC, Ivy SP, Matulonis UA. Combination cediranib and olaparib versus olaparib alone for women with recurrent platinum-sensitive ovarian cancer: a randomised phase 2 study. Lancet Oncol. 2014 Oct;15(11):1207-14. doi: 10.1016/S1470-2045(14)70391-2. Epub 2014 Sep 10. PMID 25218906
- [Derived] Liu JF, Tolaney SM, Birrer M, Fleming GF, Buss MK, Dahlberg SE, Lee H, Whalen C, Tyburski K, Winer E, Ivy P, Matulonis UA. A Phase 1 trial of the poly(ADP-ribose) polymerase inhibitor olaparib (AZD2281) in combination with the anti-angiogenic cediranib (AZD2171) in recurrent epithelial ovarian or triple-negative breast cancer. Eur J Cancer. 2013 Sep;49(14):2972-8. doi: 10.1016/j.ejca.2013.05.020. Epub 2013 Jun 27. PMID 23810467

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 0 (20mg Ced+100mg Olap); Dose Level 1 (20mg Ced + 200mg Olap); Dose Level 2 (30mg Ced + 200mg Olap); Dose Level 3 (30mg Ced + 400mg Olap); Expansion Cohort at MTD: Assess the maximum tolerated dose (MTD) of cediranib in combination with olaparib in the treatment of recurrent ovarian, fallopian tube, or peritoneal cancer or metastatic triple-negative breast cancer.
- Phase 2 - Olaparib Alone: Phase 2 - a total of 46 patients were randomized to receive olaparib alone.
- Phase 2 - Cediranib/Olaparib: Phase 2 - a total of 44 patients were randomized to receive cediranib and olaparib.
- Phase 1-T Dose Level 0-TA: Cediranib 30mg PO daily; Olaparib (tablet) 150mg PO BID
- Phase 1-T Dose Level 1-TA: Cediranib 30mg PO daily; Olaparib (tablet) 200mg PO BID
- Phase 1-T Dose Level 2-TA: Cediranib 30mg PO daily; Olaparib (tablet) 250mg PO BID
- Phase 1-T Dose Level 0-TB: Cediranib 20mg PO daily; Olaparib (tablet) 200mg PO BID
- Phase 1-T Dose Level 1-TB: Cediranib 20mg PO daily; Olaparib (tablet) 250 mg PO BID
- Phase 1-T Dose Level 2-TB: Cediranib 20mg PO daily; Olaparib (tablet) 300mg PO BID
- Phase 1-T PKOlap Expansion: Cediranib 30mg PO daily; Olaparib (tablet) 200mg BID; 7-day lead-in of single-agent olaparib
- Phase 1-T PKCed Expansion: Cediranib 30mg PO daily; Olaparib (tablet) 200mg BID; 7-day lead-in of single agent cediranib
Period: Phase 1 Dose Level 0
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1 Dose Level 1
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1 Dose Level 2
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1 Dose Level 3
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Expansion at Maximum Tolerated Dose
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 0 | 0 | 0 | 0 | 46 | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 46 | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1-T Dose Level 0-TA
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1-T Dose Level 1-TA
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1-T Dose Level 2-TA
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1-T Dose Level 0-TB
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1-T Dose Level 1-TB
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1-T Dose Level 2-TB
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1-T PKOlap Expansion
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1-T PKCed Expansion
Arm/Group | Dose Level 0 (20mg Ced+100mg Olap) | Dose Level 1 (20mg Ced + 200mg Olap) | Dose Level 2 (30mg Ced + 200mg Olap) | Dose Level 3 (30mg Ced + 400mg Olap) | Expansion Cohort at MTD | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Phase 1 was composed of 20 ovarian patients & 8 breast patients Phase 2 was composed of 90 ovarian patients Phase 1-T was composed of 37 ovarian patients
Groups:
- Phase 1 Dose Level 0 (3 Participants); Phase 1 Dose Level 1 (3 Participants); Phase 1 Dose Level 2 (7 Participants); Phase 1 Dose Level 3 (6 Participants); Phase 1 Expansion at MTD (9 Participants): Assess the maximum tolerated dose (MTD) of cediranib in combination with olaparib in the treatment of recurrent ovarian, fallopian tube, or peritoneal cancer or metastatic triple-negative breast cancer.
  This was an open-label, phase 1, dose-escalation trial performed at two participating institutions evaluating increasing doses of once daily cediranib and twice daily olaparib administered continuously in 28-day cycles. Cediranib was administered as 10 and 15 mg tablets and olaparib as 50 mg capsules. The primary objectives were to determine the dose limiting toxicities (DLT) and maximum tolerated dose (MTD) of this combination. Secondary objectives included assessment of treatment-related toxicities and preliminary assessment of clinical activity as measured by response rate, clinical benefit rate (CBR) and progression-free survival (PFS), defined as time from initiation of therapy to disease progression or death from any cause.
- Phase 2 - Olaparib Alone: Assess the efficacy (as measured by progression-free survival (PFS) ) of olaparib alone in recurrent grade 2 or 3 platinum-sensitive papillary-serous or endometrioid ovarian, fallopian tube, or peritoneal cancer.
- Phase 2 - Cediranib/Olaparib: Assess the efficacy (as measured by progression-free survival (PFS) ) of the combination of cediranib and olaparib in recurrent grade 2 or 3 platinum-sensitive papillary-serous or endometrioid ovarian, fallopian tube, or peritoneal cancer.
- Phase 1-T Dose Level 2-TA: Cediranib 30mg PO daily; Olaparib (tablet) 250mgPO BID
- Phase 1-T Dose Level 1-TB: Cediranib 20mg PO daily; Olaparib (tablet) 250mg PO BID
- Phase 1-T PKOlap Expansion: Cediranib 30mg PO daily; Olaparib (tablet) 200mg PO BID; 7-day lead-in of single-agent olaparib
- Phase 1-T PKCed Expansion: Cediranib 30mg PO daily; Olaparib (tablet) 200mg PO BID; 7-day lead-in of single-agent cediranib
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 0 (3 Participants) | Phase 1 Dose Level 1 (3 Participants) | Phase 1 Dose Level 2 (7 Participants) | Phase 1 Dose Level 3 (6 Participants) | Phase 1 Expansion at MTD (9 Participants) | Phase 2 - Olaparib Alone | Phase 2 - Cediranib/Olaparib | Phase 1-T Dose Level 0-TA | Phase 1-T Dose Level 1-TA | Phase 1-T Dose Level 2-TA | Phase 1-T Dose Level 0-TB | Phase 1-T Dose Level 1-TB | Phase 1-T Dose Level 2-TB | Phase 1-T PKOlap Expansion | Phase 1-T PKCed Expansion | Total
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 9 | 46 | 44 | 3 | 6 | 3 | 3 | 3 | 6 | 6 | 7 | 155
Age, Continuous [Mean (Full Range); unit: years] | 49 [39 to 69] | 59 [53 to 63] | 57 [36 to 71] | 56 [46 to 68] | 57 [45 to 69] | 58.1 [32.7 to 81.9] | 57.8 [41.9 to 85.6] | 55.6 [45.5 to 63.3] | 61.5 [38.3 to 71.7] | 58.7 [47.7 to 79.9] | 57.8 [48.6 to 70.1] | 59.0 [54.9 to 63.8] | 59.8 [40.3 to 76.6] | 58.7 [47.0 to 69.6] | 54.5 [41.5 to 66.9] | 57.7 [32.7 to 85.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 7 | 6 | 9 | 46 | 44 | 3 | 6 | 3 | 3 | 3 | 6 | 6 | 7 | 155
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 7 | 5 | 9 | 44 | 43 | 3 | 5 | 3 | 3 | 3 | 6 | 5 | 7 | 149
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5
  White | 3 | 3 | 6 | 4 | 9 | 42 | 43 | 3 | 5 | 2 | 2 | 3 | 4 | 6 | 6 | 141
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 7 | 6 | 9 | 46 | 44 | 3 | 6 | 3 | 3 | 3 | 6 | 6 | 7 | 155
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status
  0. Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 2 | 0 | 2 | 1 | 4 | 34 | 31 | 2 | 6 | 2 | 3 | 2 | 4 | 5 | 7 | 105
    1 | 1 | 3 | 5 | 5 | 5 | 12 | 13 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 50
Diagnosis [Count of Participants; unit: Participants]
  Ovarian | 2 | 2 | 5 | 4 | 7 | 46 | 44 | 3 | 6 | 3 | 3 | 3 | 6 | 6 | 7 | 147
  Breast | 1 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
BRCA Status [Count of Participants; unit: Participants]
  Mutation carrier | 1 | 2 | 5 | 3 | 4 | 24 | 23 | 2 | 2 | 2 | 0 | 1 | 3 | 2 | 1 | 75
  Wild-type | 2 | 0 | 0 | 0 | 2 | 11 | 12 | 1 | 4 | 1 | 3 | 2 | 2 | 3 | 5 | 48
  Unknown | 0 | 1 | 2 | 3 | 3 | 11 | 9 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 32
Number of prior regimens (median; Phase 1) [Median (Full Range); unit: number of prior regimens] — Population: Participants were assessed according to diagnosis.
  number of prior regimens
    Ovarian: number analyzed (Participants) | 2 | 2 | 5 | 4 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20
    Ovarian | 3.5 [2 to 5] | 6.5 [1 to 12] | 2 [1 to 5] | 2 [1 to 4] | 1 [1 to 5] |  |  |  |  |  |  |  |  |  |  | 2 [1 to 12]
    Breast: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
    Breast | 3 [3 to 3] | 3 [3 to 3] | 5 [4 to 6] | 2 [2 to 2] | 2.5 [2 to 3] |  |  |  |  |  |  |  |  |  |  | 3 [2 to 6]
Number of Prior Lines (Phase 2 and 1-T) [Count of Participants; unit: Participants] — Population: Number of Prior Lines was captured as displayed for Phase 2 and Phase 1-T cohorts.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 46 | 44 | 3 | 6 | 3 | 3 | 3 | 6 | 6 | 7 | 127
    1 |  |  |  |  |  | 17 | 26 | 1 | 3 | 1 | 1 | 0 | 2 | 2 | 2 | 55
    2 |  |  |  |  |  | 18 | 10 | 1 | 1 | 1 | 0 | 0 | 3 | 1 | 5 | 40
    3 or More |  |  |  |  |  | 11 | 8 | 1 | 2 | 1 | 2 | 3 | 1 | 3 | 0 | 32
Platinum-sensitivity (ovarian patients only) [Count of Participants; unit: Participants] — Population: Platinum-sensitivity is reported only for the Ovarian cohort
  Participants
    number analyzed (Participants) | 2 | 2 | 5 | 4 | 7 | 46 | 44 | 3 | 6 | 3 | 3 | 3 | 6 | 6 | 7 | 147
    Platinum-sensitive | 0 | 2 | 4 | 4 | 4 | 46 | 44 | 0 | 3 | 2 | 1 | 1 | 2 | 2 | 4 | 119
    Platinum-resistant | 2 | 0 | 1 | 0 | 3 | 0 | 0 | 3 | 3 | 1 | 2 | 2 | 4 | 4 | 3 | 28
Histology (ovarian patients only; Phase 1 and Phase 2) [Count of Participants; unit: Participants] — Population: Histologic subtype only applies to the Ovarian cohort
  Participants
    number analyzed (Participants) | 2 | 2 | 5 | 4 | 7 | 46 | 44 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 113
    Papillary-serous | 2 | 2 | 3 | 3 | 6 | 40 | 41 | 2 |  |  |  |  |  |  |  | 99
    Endometrioid | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 |  |  |  |  |  |  |  | 6
    Mixed | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 |  |  |  |  |  |  |  | 4
    Other | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 |  |  |  |  |  |  |  | 4
Histology (Phase 1-T) [Count of Participants; unit: Participants] — Population: Histologic sub-types were captured/displayed differently between phases in this trial. The histologic subtypes in this table refer to those captured/displayed for Phase 1-T participants.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 3 | 3 | 6 | 6 | 7 | 37
    Serous |  |  |  |  |  |  |  | 2 | 5 | 2 | 3 | 2 | 4 | 4 | 6 | 28
    Endometrioid |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
    Clear Cell |  |  |  |  |  |  |  | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3
    Other/Unknown |  |  |  |  |  |  |  | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities of Cediranib Maleate in Combination With Olaparib (Phase I)
Description: Was determined using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: At 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Level 0; Level 1; Level 2; Level 3: Assess the maximum tolerated dose (MTD) of cediranib in combination with olaparib in the treatment of recurrent ovarian, fallopian tube, or peritoneal cancer or metastatic triple-negative breast cancer.
Arm/Group | Level 0 | Level 1 | Level 2 | Level 3
Number analyzed (Participants) | 3 | 3 | 7 | 6
Participants | 0 | 0 | 0 | 2
Statistical Analysis 1: Comparison: Level 0 vs Level 1 vs Level 2 vs Level 3; Test type: Other; Maximum Tolerated Dose (mg) = 30 — Cediranib
Statistical Analysis 2: Comparison: Level 0 vs Level 1 vs Level 2 vs Level 3; Test type: Other; Maximum Tolerated Dose (mg BID) = 200 — Olaparib

2. Primary Outcome: The Maximum Tolerated Dose (MTD) of Cediranib in Combination With Olaparib in the Treatment of Recurrent Ovarian, Fallopian Tube, or Peritoneal Cancer or Metastatic Triple-negative Breast Cancer (Phase I)
Description: This trial employed a 3+3 design, escalating on 0/3 or 1/6 DLT, and de-escalating if 2 DLTs were encountered. The MTD (maximum tolerated dose) was the dose at which no more than 1 patient developed a dose-limiting toxicity (DLT) when at least 6 patients had been treated.
Time Frame: At 28 Days
Measure: Number; unit: mg
Groups:
- All Phase 1 Participants (28 Participants): All Phase 1 participants who received at least 1 dose of olaparib and cediranib.
Arm/Group | All Phase 1 Participants (28 Participants)
Number analyzed (Participants) | 28
mg
  Cediranib PO daily | 30
  Olaparib PO BID | 200

3. Primary Outcome: Progression-free Survival (PFS) at the Maximum Tolerated Dose/Recommended Phase 2 Dose of Cediranib Maleate With Olaparib Compared to That of Olaparib Alone (Phase II)
Description: Evaluated by Kaplan-Meier analysis and log-rank test for between group comparison, and median survival times reported.
  PFS is defined as time from randomization to investigator-assessed radiographic progression by RECIST 1.1 criteria or death.
  Patients alive without evidence of progression were censored at the last disease assessment.
Time Frame: Time from start of treatment to time of objective disease progression, assessed up to 5 years
Population: Platinum-sensitive recurrent grade 2 or 3 platinum-sensitive papillary-serous or endometrioid ovarian, fallopian tube, or peritoneal cancer.
Measure: Median (Full Range); unit: months
Groups:
- Phase 2 - Olaparib Alone (46 Participants): Assess the efficacy (as measured by progression-free survival (PFS) ) of olaparib alone in recurrent grade 2 or 3 platinum-sensitive papillary-serous or endometrioid ovarian, fallopian tube, or peritoneal cancer.
- Phase 2 - Cediranib/Olaparib (44 Participants): Assess the efficacy (as measured by progression-free survival (PFS) ) of the combination of cediranib and olaparib in recurrent grade 2 or 3 platinum-sensitive papillary-serous or endometrioid ovarian, fallopian tube, or peritoneal cancer.
Arm/Group | Phase 2 - Olaparib Alone (46 Participants) | Phase 2 - Cediranib/Olaparib (44 Participants)
Number analyzed (Participants) | 46 | 44
months | 8.2 [1 to 49] | 16.5 [4 to 60]
Statistical Analysis 1: Comparison: Phase 2 - Olaparib Alone (46 Participants) vs Phase 2 - Cediranib/Olaparib (44 Participants); Test type: Superiority; p = 0.006, Kaplan-Meier Plot; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.30 to 0.83]

4. Primary Outcome: The Maximum Tolerated Dose (MTD) of Cediranib in Combination With Olaparib Tablet Formulation in the Treatment of Recurrent Ovarian, Fallopian Tube, or Peritoneal Cancer (Phase I-T).
Description: The Phase 1-T component of this trial employed a 3+3 design, escalating on 0/3 or 1/6 DLT, and de-escalating if 2 DLTs were encountered. The MTD (maximum tolerated dose) was the dose at which no more than 1 patient developed a DLT when at least 6 patients had been treated.
Time Frame: At 28 days
Measure: Number; unit: mg
Groups:
- All Phase 1-T Participants: All Phase 1-T participants who received protocol treatment.
Arm/Group | All Phase 1-T Participants
Number analyzed (Participants) | 37
mg
  Cediranib PO daily | 30
  Olaparib (tablet) PO BID | 200

5. Secondary Outcome: Number of Participants With Treatment-related Toxicities of the Combination of Cediranib Maleate and Olaparib (Phase I)
Description: Will be determined using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0, study-related adverse events observed in >10% of participants (n=28).
Time Frame: Adverse Events monitored for 3 years, mortality assessed up to 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Tumor Response Rate (Objective Response Rate) Defined by Response Evaluation Criteria in Solid Tumors Criteria (Phase II)
Description: The response rates are compared by an exact test and 95% confidence intervals will also be reported.
  Objective response rate (ORR) is defined as the best confirmed RECIST response, ORR is defined as the number of participants with CR, PR or SD.
Time Frame: Up to 5 years
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival (Phase II)
Description: Will be evaluated by Kaplan-Meier analysis and log-rank test for between-group comparison, and median survival time will be reported.
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Secondary Outcome: Number of Participants With Treatment-related Toxicities of the Combination of Cediranib and Olaparib (Tablet Formulation) in the Treatment of Recurrent Ovarian, Fallopian Tube, or Peritoneal Cancer (Phase I-T).
Description: Will be determined using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. This outcome reports treatment-related adverse events that occurred in at least 10% of participants.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events monitored for 3 years, mortality assessed up to 5 years
Groups:
- Phase I Dose Level 0: Participants received cediranib 20 mg daily and olaparib 100 mg twice daily.
  Cediranib was administered as 10 and 15 mg tablets and olaparib as 50 mg capsules.
- Phase I Dose Level 1: Participants received cediranib 20 mg daily and olaparib 200 mg twice daily.
  Cediranib was administered as 10 and 15 mg tablets and olaparib as 50 mg capsules.
- Phase I Dose Level 2; Phase I Expansion Cohort at MTD: Participants received cediranib 30 mg daily and olaparib 200 mg twice daily.
  Cediranib was administered as 10 and 15 mg tablets and olaparib as 50 mg capsules.
- Phase I Dose Level 3: Participants received cediranib 30 mg daily and olaparib 400 mg twice daily.
  Cediranib was administered as 10 and 15 mg tablets and olaparib as 50 mg capsules.
- Phase II Olaparib Alone: Participants received olaparib capsule monotherapy 400 mg orally twice daily.
- Phase II Cediranib/Olaparib: Participants received a previously established recommended Phase 2 dose of cediranib 30 mg orally daily with olaparib capsules 200 mg orally twice daily.
- Phase I-T Dose Level 0-TA: Participants received 30 mg cediranib daily with olaparib tablets at 150 mg twice daily.
- Phase I-T Dose Level 1-TA; Phase I-T Dose Level 1-TPKCed; Phase I-T Dose Level 1-TPKOlap: Participants received 30 mg cediranib daily with olaparib tablets at 200 mg twice daily.
- Phase I-T Dose Level 2-TA: Participants received 30 mg cediranib daily with olaparib tablets at 250 mg twice daily.
- Phase I-T Dose Level 0-TB: Participants received 20 mg cediranib daily with olaparib tablets at 200 mg twice daily.
- Phase I-T Dose Level 1-TB: Participants received 20 mg cediranib daily with olaparib tablets at 250 mg twice daily.
- Phase I-T Dose Level 2-TB: Participants received 20 mg cediranib daily with olaparib tablets at 300 mg twice daily.
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase I Dose Level 3 | Phase I Expansion Cohort at MTD | Phase II Olaparib Alone | Phase II Cediranib/Olaparib | Phase I-T Dose Level 0-TA | Phase I-T Dose Level 1-TA | Phase I-T Dose Level 1-TPKCed | Phase I-T Dose Level 1-TPKOlap | Phase I-T Dose Level 2-TA | Phase I-T Dose Level 0-TB | Phase I-T Dose Level 1-TB | Phase I-T Dose Level 2-TB
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 6/7 | 6/6 | 7/9 | 29/46 | 26/44 | 1/3 | 2/6 | 2/7 | 3/6 | 1/3 | 1/3 | 2/3 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 0/7 | 2/6 | 0/9 | 2/46 | 3/44 | 0/3 | 0/6 | 1/7 | 0/6 | 1/3 | 0/3 | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 7/7 | 6/6 | 9/9 | 45/46 | 44/44 | 3/3 | 6/6 | 7/7 | 6/6 | 3/3 | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 0 (N=3) | Phase I Dose Level 1 (N=3) | Phase I Dose Level 2 (N=7) | Phase I Dose Level 3 (N=6) | Phase I Expansion Cohort at MTD (N=9) | Phase II Olaparib Alone (N=46) | Phase II Cediranib/Olaparib (N=44) | Phase I-T Dose Level 0-TA (N=3) | Phase I-T Dose Level 1-TA (N=6) | Phase I-T Dose Level 1-TPKCed (N=7) | Phase I-T Dose Level 1-TPKOlap (N=6) | Phase I-T Dose Level 2-TA (N=3) | Phase I-T Dose Level 0-TB (N=3) | Phase I-T Dose Level 1-TB (N=3) | Phase I-T Dose Level 2-TB (N=6)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Serum amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 0 (N=3) | Phase I Dose Level 1 (N=3) | Phase I Dose Level 2 (N=7) | Phase I Dose Level 3 (N=6) | Phase I Expansion Cohort at MTD (N=9) | Phase II Olaparib Alone (N=46) | Phase II Cediranib/Olaparib (N=44) | Phase I-T Dose Level 0-TA (N=3) | Phase I-T Dose Level 1-TA (N=6) | Phase I-T Dose Level 1-TPKCed (N=7) | Phase I-T Dose Level 1-TPKOlap (N=6) | Phase I-T Dose Level 2-TA (N=3) | Phase I-T Dose Level 0-TB (N=3) | Phase I-T Dose Level 1-TB (N=3) | Phase I-T Dose Level 2-TB (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 4 | 15 | 20 | 2 | 2 | 3 | 4 | 2 | 3 | 3 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 3 | 1 | 4 | 6 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 3 | 1 | 0 | 5 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 4
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 0 | 3 | 6 | 14 | 1 | 1 | 1 | 0 | 0 | 3 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 6 | 11 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 2 | 0 | 7 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 5 | 7 | 1 | 1 | 3 | 0 | 0 | 1 | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 8 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood and lymphatic system disorders - Other, NOS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac disorders - Other, NOS (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholesterol high (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Concentration impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 5 | 1 | 2 | 15 | 18 | 0 | 3 | 2 | 2 | 1 | 2 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 3 | 11 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2
Creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 3 | 6 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 6 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 6 | 5 | 9 | 14 | 41 | 3 | 6 | 5 | 5 | 2 | 3 | 2 | 5
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 2 | 6 | 10 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 6 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Dysesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 5 | 6 | 0 | 1 | 2 | 0 | 2 | 1 | 2 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 10 | 11 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 2 | 3 | 11 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 1 | 0 | 1 | 6 | 9 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, NOS (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 6 | 6 | 9 | 36 | 40 | 3 | 6 | 5 | 6 | 3 | 3 | 3 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 8 | 0 | 3 | 0 | 2 | 1 | 0 | 1 | 0
Gastrointestinal disorders - Other, NOS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 3 | 8 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
General disorders and administration site conditions - Other, NOS (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gum infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 3 | 2 | 4 | 9 | 24 | 1 | 3 | 3 | 3 | 1 | 1 | 2 | 3
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1 | 1 | 0 | 12 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 1 | 0 | 2 | 4 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 4 | 3 | 3 | 8 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 3 | 4 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 8 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 1 | 1 | 11 | 10 | 1 | 2 | 3 | 1 | 0 | 1 | 1 | 4
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 1 | 3 | 11 | 1 | 3 | 4 | 1 | 0 | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2 | 2 | 2 | 3 | 0 | 8 | 0 | 3 | 2 | 1 | 0 | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, NOS (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Injury, poisoning and procedural complications - Other, NOS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INR increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 2 | 3 | 8 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, NOS (Investigations) | 0 | 0 | 1 | 3 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 3 | 0 | 4 | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, NOS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 9 | 2 | 2 | 0 | 1 | 1 | 2 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, NOS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 5 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 7 | 0 | 3 | 0 | 3 | 0 | 1 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 4 | 4 | 7 | 36 | 35 | 3 | 5 | 4 | 5 | 1 | 3 | 3 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorders - Other, NOS (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 2 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 2 | 3 | 7 | 8 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 4 | 6 | 11 | 2 | 1 | 2 | 3 | 0 | 1 | 1 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 8 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 0 | 3 | 3 | 11 | 16 | 2 | 5 | 3 | 3 | 2 | 1 | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0
Psychiatric disorders - Other, NOS (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, NOS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus pain (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 3 | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, NOS (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 4 | 4 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, NOS (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 4 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Transient ischemic attacks (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 6 | 9 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 5 | 6 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 4
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular disorders - Other, NOS (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 3 | 3 | 14 | 11 | 3 | 3 | 3 | 2 | 1 | 1 | 1 | 4
Weight gain (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 2 | 1 | 1 | 0 | 12 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
White blood cell decreased (Investigations) | 1 | 1 | 2 | 2 | 2 | 6 | 7 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT01116648/Prot_SAP_000.pdf